CLINICAL TRIAL: NCT07010783
Title: Investigation of Respiratory Functions, Inspiratory Muscle Strength, Physical Fitness and Aerobic Capacity in Patients With Parkinson's Disease
Brief Title: Respiratory Functions in Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: Ankara University (Other)
Collaborators: Hacettepe University (Other); Atılım University (Other)
Responsible Party: Principal Investigator, Büşra Seçkinoğulları Korkusuz, Principal Investigator, Ankara University
Other Study IDs: E-59394181-604.01-112206
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Early Stage Patients with Parkinson's Disease: According to the Modified Hoehn and Yahr Scale (MHÖ), patients with a score below 2.5
- Advanced Stage Patients with Parkinson's Disease: According to the Modified Hoehn and Yahr Scale (MHÖ), patients with 2.5 and above
- Control Group: Healthy individuals with similar demographic characteristics

SUMMARY:
The aim is to examine respiratory functions, inspiratory muscle strength, respiratory function, physical fitness and aerobic capacity in Parkinson's disease patients. Individuals between the ages of 50-80 who have been diagnosed with Parkinson's disease by a neurologist and healthy individuals with similar demographic characteristics will be included in the study as a control group. In addition, patients will be divided into three groups as above and below 2.5 and healthy controls according to the Modified Hoehn and Yahr Scale. Demographic information of the individuals will be recorded and clinical evaluations will be made. The staging of Parkinson's patients will be done with the Modified Hoehn and Yahr Scale, and the severity of the disease will be done with the Unified Parkinson's Disease Rating Scale. The inspiratory muscle strength of the individuals will be evaluated with the PowerBreath K5, respiratory functions with the Pulmonary Function Test device, and physical fitness and aerobic capacity with the Senior Fitness Test.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 to 80
* Mini Mental State Examination score of 24 to 30
* Diagnosed with Parkinson's Disease by a neurologist

Exclusion Criteria:

* Sözlü iletişim kuramama
* Yürüme yardımcısı kullanıma
* Ciddi görme bozukluğu, ek nörolojik bozuklukları ve/veya konjestif kalp yetmezliği olan yaşlılar
* Egzersiz yapılması tavsiye edilmeyen yaşlı yetişkinler.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease who came to the neurology outpatient clinic for routine examination and who met the appropriate inclusion criteria and healthy individuals with similar demographic characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Inspiratory Muscle Strength Measurement | Baseline
  In this study, the inspiratory muscle strength of the participants will be measured using the Power Breath device.
Unified Parkinson's Disease Rating Scale | Baseline
  This scale will evaluate the severity and stage of the participants' Parkinson's disease.
Evaluation of Respiratory Functions | Baseline
  Participants' respiratory functions will be evaluated using a standard respiratory function test device.
Senior Fitness Test | Baseline
  The physical fitness levels of the participants will be evaluated using the Senior Fitness Test.

CONTACTS AND LOCATIONS:
Overall Officials: Süleyman Korkusuz, PhD, Study Chair — Atılım University; Ayla Fil Balkan, Assoc Prof, Study Chair — Hacettepe University; Gül Yalçın Çakmaklı, Assoc Prof, Study Chair — Hacettepe University; Neslihan Durutürk, Prof.Dr, Study Chair — Baskent University
Locations (1):
- Atılım University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shill H, Stacy M. Respiratory function in Parkinson's disease. Clin Neurosci. 1998;5(2):131-5. PMID 10785839
- [Result] Morris ME, Iansek R, Matyas TA, Summers JJ. Ability to modulate walking cadence remains intact in Parkinson's disease. J Neurol Neurosurg Psychiatry. 1994 Dec;57(12):1532-4. doi: 10.1136/jnnp.57.12.1532. PMID 7798986